CLINICAL TRIAL: NCT05954585
Title: The Development of a Family Navigator Intervention and Prevention Protocol to Reduce Risk of Suicide and Self-injurious Behavior for Youth Aged 8 to 14 Years
Brief Title: Family Navigator Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Graduated off COBRE grant
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Mary Kathryn Cancilliere, Research Scientist / Assistant Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RIH.100
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Treatment as Usual; Family Navigator
Keywords: emergency department, suicide, youth, family navigator
MeSH Terms: conditions — Emergencies; Suicide | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person conducting follow-up assessments will be masked as to the intervention assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Emergency department treatment as usual
  Interventions: Behavioral: Treatment as usual
- Family Navigator (Experimental): Follow provision provided by a Family Navigator for the length of the treatment or until youth attends community-based mental health care
  Interventions: Behavioral: Family Navigator

INTERVENTIONS:
Behavioral: Treatment as usual — Emergency department treatment as usual
  Arms: Treatment as usual
Behavioral: Family Navigator — Family Navigator will speak with families about individual and systemic issues for linkage to mental health care biweekly for 3 months or until the youth's first mental health appt has been attended, whichever comes first.
  Arms: Family Navigator

SUMMARY:
This study will develop and examine the feasibility and acceptability of a family navigator protocol while leveraging digital health communication. It will employ an ecological model within a socio-cultural theoretic framework of mental health service disparities and barriers to treatment.

DETAILED DESCRIPTION:
The purpose of this study is to develop and pilot a Family Navigator intervention with technology-enhanced information sharing for families with youth (80 youth-caregiver dyads) who were discharged from the emergency after an admission for SSIB. This novel intervention aims to reduce suicidal and non-suicidal self-injurious behavior risk and prevalence rates by way of increasing attendance to community-based mental health services for youth aged 10 to 14.

ELIGIBILITY:
Inclusion Criteria:

* youth 10 to 14 years old living at home with legal guardian/caregiver

Exclusion Criteria:

* presentation including psychosis, sexual assault, or child abuse,
* are in police or child protective services' custody,
* are unable to assent due to severity of illness or developmental disabilities, >cannot communicate in English or Spanish, or
* if no caregiver or legal guardian is able to provide consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Mental Health Services | 6 months
  adapted CASA

SECONDARY OUTCOMES:
Suicidal ideation | 6 months
  Suicidal Ideation Questionnaire
Suicidal behavior | 6 months
  Suicidal Ideation Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kathryn Cancilliere, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided